CLINICAL TRIAL: NCT04573530
Title: We Walk Plus Study: A Walking Program Using Physical Activity Monitors and Social Networking for Older Adults With Intellectual Disabilities
Brief Title: We Walk Plus Study for Older Adults With Intellectual Disabilities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kueifang Hsieh, Research Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2020-1140
Record Dates: First submitted 2020-09-14; First posted 2020-10-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability
Keywords: physical activity; walking; older adults with an intellectual disability
MeSH Terms: conditions — Intellectual Disability; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- We Walk Plus Intervention (Experimental): The intervention group will receive a Fitbit, SMS and will be assigned to a private Fitbit community (4-5 participants per group) for 12 weeks. During the intervention, participants will receive weekly personalized SMS on their mobile phones including encouraging messages, reminders, and tips to increase steps, and weekly step goals. The investigators will use a secure, web-based platform, iCardia, to support continuous real-time remote monitoring of activity data from Fitbit devices and personalized communication via SMS based on incoming data. The investigators will set up the Fitbit networking settings on participants' phones to give notifications when there are posts to this group. Individual goals and a weekly team goal of steps will be set up by the research team. Each member will be awarded a badge upon reaching each individual's weekly goal. Teams will also be awarded badges when all team members reach their individual weekly goals.
  Interventions: Behavioral: We Walk Plus Intervention
- Attention control group (No Intervention): The attention control group will also receive a Fitbit and will be asked to continue with normal daily activities. During the initial in-person session, they will receive the same PA recommendations as the intervention group to walk at least 30 minutes for 5 days or more a week or 10,000 steps a day. However, a plan for improving PA will not be discussed.

INTERVENTIONS:
Behavioral: We Walk Plus Intervention — The frequency and content of weekly personalized SMS are based on each participant's preference. Prior to implementation of intervention, the investigators will conduct focus groups to learn participants' social network activities and preferences, strategies that can be used to encourage engagement via a private Fitbit community network.
  Arms: We Walk Plus Intervention

SUMMARY:
Determine the feasibility and acceptability of We Walk Plus intervention to promote physical activity and improve cognition for older adults with intellectual disabilities (ID).

DETAILED DESCRIPTION:
We Walk Plus study consists of: (1) a user friendly physical activity tracker (i.e., Fitbit Charge HR ); (2) user-centered social networking (e.g., Fitbit community); and (3) the iCardia platform for monitoring daily Fitbit physical activity and wear time and sending personalized text-messages targeting physical activity and self-efficacy. The specific aims of this two-arm RCT pilot are to: 1) assess the feasibility and acceptability of the We Walk Plus intervention and 2) explore the preliminary efficacy of We Walk Plus on physical activity and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with mild or moderate intellectual disabilities;
* ages 35-60;
* able to speak, read English and willing to provide consent to enroll;
* able to follow instructions and walk, physically inactive;
* willing to receive SMS, wear Fitbit throughout the study;
* living with family or in a community residence;
* support persons are willing to assist participants to ensure the Fitbit functions properly.

Exclusion Criteria:

* Inability to follow instructions;
* diagnosis of coronary disease or uncontrolled hypertension, smokers, physically active;
* participating in a health promotion program;
* having mental illness or behavior problems;
* support persons unable or unwilling to assist participants with Fitbit devices, if needed.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 12 weeks
  daily steps

SECONDARY OUTCOMES:
Cardiovascular fitness | 12 weeks
  modified six-minute walk test
Self-efficacy to physical activity | 12 weeks
  Physical Activity Self-efficacy/Social Support scale will be used to assess confidence to perform physical activity
Attention & executive function | 12 weeks
  Flanker Inhibitory Control and Attention Test -a standard test from the NIH toolbox which has been adapted and validated for individuals with ID to assess one's limited capacities to deal with an abundance of environmental stimulation.
Working memory | 12 weeks
  List Sorting Working Memory Test-a standard test from the NIH toolbox which has been adapted and validated for individuals with ID to assess the ability to store information.
Executive function | 12 weeks
  Dimensional Change Card Sort Test -a standard test from the NIH toolbox which has been adapted and validated for individuals with ID to assess one's capacity to plan, organize, and monitor the executive of behaviors.
Processing speed | 12 weeks
  Pattern Comparison Processing Speed Test- a standard test from the NIH toolbox which has been adapted and validated for individuals with ID to assess the amount of information that can be processed within a certain unit of time.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Trinity Services Inc., New Lenox, Illinois